CLINICAL TRIAL: NCT06389682
Title: Pharmacokinetics, Biodistribution, Radiation Dose and Safety Study of a Single Dose of Gallium [68Ga]-NYM005 Injection Prepared by Kit for the Preparation of the 68Ga-NYM005 Injection in Patients With Metastatic Clear Cell Renal Carcinoma.
Brief Title: Pharmacokinetics, Biodistribution, Radiation Dose and Safety Study of 68Ga-NYM005 in Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Norroy Bioscience Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-2023-02
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Clear Cell Renal Cell Carcinoma Metastatic
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-NYM005 injection (Experimental)
  Interventions: Drug: 68Ga-NYM005 injection

INTERVENTIONS:
Drug: 68Ga-NYM005 injection — he radiation dose is about 2-7 mCi for a single patient.Using a syringe to withdraw 68Ga-NYM005 injection, the dose will be administered via an intravenous injection and the injection time will be about 45-60 seconds.

SUMMARY:
68Ga-NYM005 is a CAIX-targeting small-molecular radiotracer for PET/CT imaging of clear cell renal cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed metastatic renal clear cell carcinoma;
2. Age range from 18 to 75 years old (including 18 and 75 years old);
3. ECOG score of 0 or 1;
4. Expected life > 6 months;
5. GFR> 60 ml/min;
6. Women of childbearing age need to have a negative pregnancy test, and the subjects(including male subjects)agree to take effective contraceptive measures during the study period and for at least three months after the drug administration;
7. The subjects are able to maintain good communication with the researchers；understand and follow the requirements of this study and sign an informed consent form before the start of relevant research operations.

Exclusion Criteria:

1. Pregnant or lactating women, or women who plan to conceive during the study period or within three months after drug administration;
2. Known or suspected to be allergic to the investigational drug or any of its components,acetazolamide or other sulfonamides:
3. Accepting other investigational drugs upon enrollment, or within 5 biological half-lives of the drug at enrollment, or within 30 days after its last administration, whichever is longer;
4. Those who have used any radioactive therapy medication within 90 days before investigational drug administration, or have received any radioactive diagnostic medication within 3 days before investigational drug administration;
5. On VEGF TKI treatment less than 7 days before 68Ga-NYM005 PET/CT, such as sunitinib,sorafenib, cabozantinib, pazopanib, or lenvatinib, a washout of one week before 68Ga-NYM005 PET/CT is required;
6. Planned (for the period between injection of 68Ga-NYM005 and imaging) antineoplastic therapies;
7. Plan to arrange surgery and other invasive interventions within 2 days after the injection of the investigational drug;
8. Ongoing toxicity >grade l from previous standard or investigational therapies；
9. Patients with active infections during screening;
10. Those who have no guarantee of being able to lie down quietly in the examination cabin during a PET examination, or those who suffer from claustrophobia and cannot cooperate in a PET examination:
11. Other situations where the researchers believe that the subject is not suitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 5 days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Affliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Peking Union Medical College Hospital, Beijing